CLINICAL TRIAL: NCT01300962
Title: A Four Part, Phase I Dose-Escalation Study of the Combinations of Concurrent BKM120 and Capecitabine, or Concurrent BYL719 and Capecitabine, or Concurrent BKM120 and Capecitabine and Trastuzumab, or Concurrent BKM120 and Capecitabine and Lapatinib in Patients With Metastatic Breast Cancer
Brief Title: Study of BKM120 or BYL719 and Capecitabine in Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 1024; 11-0060 (Other: UNC-IRB assigned protocol number)
Record Dates: First submitted 2011-02-17; First posted 2011-02-23 (Estimated); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Metastatic Breast Cancer
Keywords: Xeloda; Capecitabine; BKM120; Lineberger Comprehensive Cancer Center; Metastatic; BYL719 Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Capecitabine; Alpelisib; Trastuzumab; Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- BYL719 ARM B (Experimental): Treatment with BYL719 and Capecitabine
  Interventions: Drug: Capecitabine; Drug: BYL719
- BKM120 ARM A (Experimental): Treatment with BKM120 and capecitabine
  Interventions: Drug: BMK120; Drug: Capecitabine
- ARM C (Experimental): BKM 120 plus capecitabine plus trastuzumab
  Interventions: Drug: BMK120; Drug: Capecitabine; Drug: Trastuzumab
- ARM D (Experimental): BKM120 plus capecitabine plus lapatinib
  Interventions: Drug: BMK120; Drug: Capecitabine; Drug: Lapatinib

INTERVENTIONS:
Drug: BMK120 — BKM120 PO 50, 80 or 100mg every day for each day of each 21 day cycle. Number of cycles: until progression of disease; unacceptable toxicity, withdrawal or death.
  Arms: ARM C; ARM D; BKM120 ARM A
Drug: Capecitabine — 875-1250mg/m2 PO BID for two weeks followed by one week rest every three week cycle. Number of cycles: until progression of disease, unacceptable toxicity, withdrawal or death.
  Other Names: Xeloda
Drug: BYL719 — BYL719 200mg PO BID for 21 days (3 weeks) in combination with capecitabine 1000 mg/m2 PO BID for 2 weeks
  Arms: BYL719 ARM B
Drug: Trastuzumab — trastuzumab infusion on day 1 of each cycle.
  Other Names: Herceptin
  Arms: ARM C
Drug: Lapatinib — lapatinib daily for 21 days in each cycle.
  Other Names: Tykerb
  Arms: ARM D

SUMMARY:
This phase I study has been designed to establish the safety, tolerability and maximum tolerated dose (MTD) of four separate regimens for patients with metastatic breast cancer: dose- escalating BKM120 when combined with capecitabine (Arm A), with capecitabine and trastuzumab (Arm C), or with capecitabine and lapatinib (Arm D) and dose- escalating BEZ235 when combined with capecitabine (Arm B).

DETAILED DESCRIPTION:
STUDY OBJECTIVES Primary Objectives

* To determine the safety, DLT, and MTD of BKM120 when administered concomitantly with capecitabine in patients with metastatic breast cancer (ARM A)
* To determine the safety, DLT, and MTD of BYL719 when administered concomitantly with capecitabine in patients with metastatic breast cancer (ARM B)
* To determine the safety, DLT, and MTD of BKM120 when administered concomitantly with capecitabine and trastuzumab in patients with metastatic breast cancer (ARM C)
* To determine the safety, DLT, and MTD of BKM120 when administered concomitantly with capecitabine and lapatinib in patients with metastatic breast cancer (ARM D)

Secondary Objectives

* To characterize the safety and tolerability of BKM120 in combination with capecitabine including acute and chronic toxicities
* To characterize the safety and tolerability ofBYL719 in combination with capecitabine including acute and chronic toxicities
* To characterize the safety and tolerability of BKM120 in combination with capecitabine and trastuzumab, including acute and chronic toxicities
* To characterize the safety and tolerability of BKM120 in combination with capecitabine and lapatinib, including acute and chronic toxicities

Exploratory Objectives

* To obtain primary, archived paraffin-embedded tissues to evaluate intrinsic breast cancer subtype (i.e., HER2, luminal B, etc.) and other important predictive biomarkers (PI3K activating mutations, pAKT, p-mTOR), and explore correlations with therapeutic response to BKM120 or BYL719 in combination with capecitabine, with or without the addition of lapatinib or trastuzumab
* To evaluate the PK profile of BKM120 with concomitant capecitabine
* To examine other signaling pathway signatures
* To examine drug effect in pre- and post-treatment core biopsy specimens (optional) from appropriate patients
* To explore patient motivators for enrolling in early phase studies through patient interview

Outline:

This study is a four-arm multi-center, open-label phase I clinical trial testing the hypothesis that the addition of BKM120 to capecitabine (ARM A); the addition of BYL719 to capecitabine (ARM B); the addition of BKM120 to capecitabine plus trastuzumab (ARM C); or the addition of BKM120 to capecitabine plus lapatinib (ARM D) will be safe and tolerable as evidenced by the DLT seen. Following screening and informed consent, treatment will be initiated with one of the following:

ARM A: BKM120 PO daily for 21 days (3 weeks) plus capecitabine PO BID for 2 weeks (no capecitabine is administered during the third week).

ARM B: BYL719 PO BID for 21 days (3 weeks) plus capecitabine PO BID for 2 weeks (no capecitabine is administered during the third week of the cycle)

ARM C: BKM120 PO daily for 21 days (3 weeks) plus capecitabine PO BID for 2 weeks (no capecitabine is administered during the third week) plus trastuzumab by intravenous infusion on Day 1

ARM D: BKM120 PO daily for 21 days (3 weeks) plus capecitabine PO BID for 2 weeks (no capecitabine is administered during the third week) plus lapatinib PO daily for 21 days.

The consents are separate documents and the patient and the study team know ahead of time which Arm is open and enrolling and can therefore focus their discussion with the patient on that ARM.

Cycles in each arm will be repeated every 3 weeks (21 days). Patients will continue on protocol-based therapy until progression, unacceptable toxicity, study withdrawal, or patient death.

ELIGIBILITY:
PATIENT ELIGIBILITY Inclusion Criteria

* Age ≥18 years (no upper age limit)
* confirmed pathologic diagnosis of breast cancer which is metastatic and for which capecitabine is a reasonable treatment option

  * ARMS C & D: Histologically confirmed HER2+ breast cancer: IHC 3+ or fluorescence in situ hybridization [FISH] amplified; by clinical assay on either primary or metastatic tumor
* Brain metastases permitted in Arms A and B if:

  * CNS-directed treatment has been given;
  * No CNS-directed therapy for the past 3 months, including glucocorticoids; AND
  * CNS disease has been clinically and radiographically stable for at least 8 weeks
* Brain metastases permitted in Arms C and D if:

  * CNS-directed treatment has been given;

    * 4 weeks interval between whole brain radiation therapy and initiation of protocol-based therapy;
    * 2 weeks interval between stereotactic radiosurgery or gamma knife (or equivalent) and initiation of protocol-based therapy;
  * CNS disease has been clinically and radiographically stable for at least 4 weeks
  * In Arm C, if patient on glucocorticoids, must be on stable (4 weeks) dose of no more than 2 mg/day of dexamethasone or equivalent.
  * In Arms B and D, no steroids are allowed.
* Measurable or non-measurable (but evaluable) disease as defined via RECIST 1.1
* No more than 4 prior chemotherapy regimens for metastatic disease for those in the dose-escalation cohorts. Prior trastuzumab and lapatinib are allowed for the HER2+ population. Once we reach the expanded RP2D cohorts, patients enrolled must have received ≤3 prior regimens

  * Patients enrolled in ARM C may remain on trastuzumab without a washout period
  * Patients enrolled in ARM D may remain on lapatinib without a washout period
* Normal organ and marrow function as defined below:

  * Absolute neutrophil count ≥1,500/μL
  * Platelets ≥100,000/μL
  * Hemoglobin ≥8.5g/dL
  * ARMs A, C, D: Total bilirubin within normal range (or ≤1.5 X upper limit of normal (ULN) if liver metastases are present); or total bilirubin ≤3.0 x ULN with direct bilirubin within normal range in patients with Gilbert Syndrome.

ARM B: Total bilirubin ≤1.5 X ULN (in patients with known Gilbert Syndrome a total bilirubin ≤3.0 x ULN with direct bilirubin ≤1.5 X ULN)

* ARMs A, C, D: AST(SGOT)/ALT(SGPT) within normal range (or ≤ 3.0X ULN if liver metastases are present) ARM B: AST(SGOT)/ALT(SGPT) ≤2.5X ULN or ≤ 5.0X ULN if liver metastases are present)
* Serum creatinine ≤1.5 X ULN OR 24-hour creatinine clearance ≥60 mL/min
* Amylase and lipase levels ≤ ULN
* Left Ventricular Ejection Fraction ≥ 50% by ECHO or MUGA

  * Total calcium (corrected for serum albumin) within normal limits (bisphosphonate use for malignant hypercalcemia control is not allowed; the use of denosumab(Xgeva®) is permitted)
  * Magnesium levels >lower limit of normal
  * ARM A: Fasting plasma glucose ≤120 mg/dL (6.7 mmol/L) ARM B: Fasting plasma glucose <140 mg/dL (7.8) mmol/L); HbA1c ≤ 8% ARMS C and D: Fasting plasma glucose ≤150 mg/dL
  * INR ≤2
  * Life expectancy ≥12 weeks
  * ECOG performance status 0-2 (Karnofsky >60%)
  * Time since the last dose of prior therapy to treat underlying malignancy:
* Cytotoxic chemotherapy or endocrine therapy: ≥ the duration of the most recent cycle of the previous regimen (with a minimum of 3 weeks for all, except 6 weeks for nitrosourea, mitomycin-C)
* Biologic therapy (e.g., antibodies): ≥4 weeks
* ≥5 X half-life of a small molecule therapeutic
* ≥4 weeks interval between whole brain radiation therapy and initiation of protocol-based therapy for ARM C or D patient with stable brain metastases;
* ≥2 weeks interval between stereotactic radiosurgery (SRS) or gamma knife (or equivalent) and initiation of protocol-based therapy for ARM C or D patient with stable brain metastases
* Patients enrolled in ARM C may remain on trastuzumab without a washout period
* Patients enrolled in ARM D may remain on lapatinib without a washout period

  -Adults of reproductive potential must be able and agree to use appropriate contraception. Double barrier contraceptives must be used throughout the trial by both sexes..
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, must use highly effective contraception during the study. Women assigned to ARMS AC and D must use highly effective contraception for 16 weeks after stopping treatment. Women assigned to ARM A must continue contraceptive measures for 4 weeks after stopping treatment. Women assigned to ARM B must continue contraceptive measures for 5 weeks after stopping treatment. The highly effective contraception is defined as either:

  * True abstinence: When this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
  * Sterilization: have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
  * Male partner sterilization (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate). For female subjects on the study, the vasectomized male partner should be the sole partner for that patient.
  * Use of a combination of any two of the following (a+b):

    1. Placement of an intrauterine device (IUD) or intrauterine system (IUS)
    2. Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel /film/cream/vaginal suppository
* For ARMs A, C and D, oral contraception (OC), injected or implanted hormonal methods are not allowed as BKM120 and potentially decreases the effectiveness of hormonal contraceptives. For ARM B, oral contraceptives, injected or implanted hormonal methods are not allowed as the sole method of contraception, as BYL719 has not been characterized with respect to its potential to interfere with the PK and/or the effectiveness of OCs.

  * Recovered from all reversible toxicities related to their previous treatment (other than alopecia) to ≤grade 1 or baseline

Exclusion Criteria:

Subjects meeting any of the exclusion criteria listed below at baseline will be excluded from study participation:

* Receiving concurrent endocrine, cytotoxic, or biologic agent(s) or within time limits specified above prior to study day 1
* Receiving any other investigational agents currently, or within time limits specified above prior to study day 1
* Received wide field radiotherapy ≤4 weeks, or SRS or gamma knife for brain metastasis ≤ 2 weeks or limited field radiation for palliation ≤2 weeks prior to starting either BYL719 or BKM120 or have not recovered from side effects of such therapy
* Have undergone major surgery ≤2 weeks prior to starting BKM120 or BYL719 or have not recovered from side effects of such therapy
* Prior treatment with treatment doses of capecitabine (prior radio-sensitizing doses of capecitabine are allowed as long as the patient did not progress on capecitabine)
* Prior treatment with a PI3K inhibitor
* Known dihydropyrimidine dehydrogenase (DPD) deficiency
* Treated with any hematopoietic colony-stimulating growth factors (e.g., G-CSF, GM-CSF) ≤2 weeks prior to starting study drug; erythropoietin or darbepoetin therapy, if initiated at least 2 weeks prior to enrollment, may be continued
* Currently receiving treatment with medication known to prolong the QT interval or inducing Torsades de Pointes and the treatment cannot either be discontinued or switched to a different medication prior to starting study drug
* Patients currently receiving chronic systemic treatment with steroids or another immunosuppressive agent; NOTE: This restriction regarding choice of glucocorticoid does not apply should patient need <2 week course of glucocorticoid for treatment of non-infectious pneumonitis during study, or if ARM C patient with brain metastases treated with glucocorticoid is enrolled. Topical applications (e.g., rash), inhaled sprays, eye drops or local injections of steroids are allowed.
* Known coagulopathies, and those who require therapeutic anticoagulation with coumarin-derivative anticoagulants
* Presence of acute or chronic liver, renal disease, or pancreatitis
* For all Arms, patients with poorly controlled diabetes mellitus, and/or with clinical signs, and/or steroid-induced diabetes mellitus; for Arm B, patients requiring insulin treatment
* History of gestational diabetes mellitus
* Known diagnosis of human immunodeficiency virus (HIV) infection
* For Arms A, C or D, patients with the following mood disorders as judged by the investigator or a psychiatrist, or as result of patient's mood assessment questionnaire:

  * Medically documented history of major depressive episode, bipolar disorder (I or II), obsessive-compulsive disorder, schizophrenia, a history of suicidal attempt or ideation, or homicidal ideation (immediate risk of doing harm to others) or patients with active severe personality disorders (defined according to DSM-IV). NOTE: for patients with psychotropic treatments ongoing at baseline, the dose and schedule should not be modified within the previous 6 weeks prior to D1 of treatment with BKM120
  * ≥ CTCAE grade 3 anxiety
  * At screening, meets the cut-off score of ≥10 in the Patient Health Questionnaire (PHQ-9) or a cut-off of ≥ 15 in the Generalized Anxiety Disorder (GAD-7) mood scale, respectively, or selects a positive response of 1, 2 or 3 to question number 9 regarding potential for suicidal thoughts in the PHQ-9 (independent of the total score of the PHQ-9) will be excluded from the study unless overruled by the psychiatric assessment

Note: The psychiatric judgment overrules the mood assessment questionnaire result/investigator's judgment.

* Not willing to avoid grapefruit, grapefruit juices, grapefruit hybrids, Seville oranges, pummelos, and exotic citrus fruits from 7 days prior to the dose of study medication and during the entire study due to potential CYP3A4 interaction with the study medication. Orange juice is allowed
* Intake of any herbal preparations or medications (e.g., including, but not limited to, Saint-Johns Wort and ginkgo biloba) and dietary supplements within 7 days prior to first dose of study drug
* For ARMS A, C and D, unable or unwilling to discontinue use of any drug known to be a strong or moderate inhibitor or inducer of CYP3A4 (prohibited inducers and inhibitors must be discontinued within 2 weeks prior to first dose of study drug) (see Appendix B); please note that co-treatment with weak inhibitors of CYP3A4 is allowed.
* Patients who received live vaccines or who have close contact with people who have received live vaccines within 7 days of day 1 of study treatment (see Appendix B)
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of BKM120 or BYL719 (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection); Patients with unresolved diarrhea will be excluded.
* Inadequately controlled hypertension (i.e. SBP >180 mmHg or DBP >100mmHg)
* Any of the following concurrent severe and/or uncontrolled medical conditions which could compromise participation in the study:

  * Left ventricular ejection fraction (LVEF) < 50% as determined by Multiple Grated acquisition (MUGA) scan or echocardiogram (ECHO)
  * ST depression or elevation of ≥1.5 mm in 2 or more leads
  * Congenital long QT syndrome
  * History or presence of ventricular arrhythmias or atrial fibrillation
  * Clinically significant resting bradycardia (<50 beats per minutes)
  * QTc >480 msec on screening ECG
  * Complete left bundle branch block
  * Right bundle branch block + left anterior hemiblock (bifascicular block)
  * Unstable angina pectoris ≤6 months prior to starting study drug
  * Acute myocardial infarction ≤6 months prior to starting study drug
  * Other clinically significant heart disease such as congestive heart failure requiring treatment (New York Heart Association [NYHA] Class III or IV)
* Other concurrent severe and/or uncontrolled concomitant medical conditions (e.g., active or uncontrolled infection) that could cause unacceptable safety risks or compromise compliance with the protocol

  * Significant symptomatic deterioration of lung function. If clinically indicated, pulmonary function tests including measures of predicted lung volumes, DLco, 02 saturation at rest on room air should be considered to exclude pneumonitis or pulmonary infiltrates
* Prior malignancy Exceptions: Subjects who have had another malignancy and have been disease-free for 3 years or subjects with a history of completely resected non-melanomatous skin carcinoma or successfully treated in situ carcinoma are eligible
* History of allergic reactions attributed to compounds of similar chemical or biologic composition of BKM120, BYL719, capecitabine (including fluorouracil), trastuzumab or lapatinib
* Pregnant or lactating women
* Patient is unable or unwilling to abide by the study protocol or cooperate fully with the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2011-08; Primary Completion 2017-02-07 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | two years
  Maximum Tolerated Dose (MTD) will be the highest does at which less than or equal to 1 out of 6 patients have experienced a dose limiting toxicity (DLT)
Dose limiting toxicity (DLT) | two years
  Dose-limiting toxicities (DLT) will be defined per NCI Common Terminology Criteria for Adverse Events version 4 (CTCAE v4)

SECONDARY OUTCOMES:
Objective Response | two years
  Objective response is measured by assessing the tumor response using Recist 1.1 criteria
Best Overall Response | two years
  The best overall response is defined as the best response achieved across all time points prior to progression (for example, a patient who has SD at first assessment, PR at second assessment, and PD on last assessment has a best overall response of PR).

CONTACTS AND LOCATIONS:
Overall Officials: Claire Dees, Principal Investigator — University of North Carolina Lineberger Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina

REFERENCES:
- See also: UNC Lineberger Comprehensive Cancer Center — http://unclineberger.org